CLINICAL TRIAL: NCT03847636
Title: Safety and Efficacy of Cryoballoon Ablation for Treatment of Sporadic and Familial Nonampullary Nonpolypoid Duodenal Adenomas (the C2D2 Trial)
Brief Title: CryoBalloon Ablation for Treatment of Duodenal Adenomas
Acronym: C2D2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00163804
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Duodenal Adenomas; Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Intervention Model Description: Non-randomized pilot study of highly selected patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Familial Adenomatous Polyposis (FAP) (Active Comparator): Individuals with duodenal adenomas (DAs) and FAP with Spigelman class 2,3 or 4, treated with cryoballoon ablation (intervention)
  Interventions: Device: CryoBalloon ablation
- Sporadic duodenal adenomas (Active Comparator): Individuals with at least 1 sporadic duodenal adenoma (DA) between 1-5 cm in maximum diameter, treated with cryoballoon ablation (intervention)
  Interventions: Device: CryoBalloon ablation

INTERVENTIONS:
Device: CryoBalloon ablation — Endoscopic cryoablation (cryogen is contained nitrous) using a CryoBalloon catheter to ablate up to 4 separate DA.

SUMMARY:
This multicenter prospective non-randomized interventional study (clinical trial) that will assess the safety and efficacy of cryoballoon ablation treatment using the C2 Cryoballoon device (Pentax Medical Corporation) as an alternative primary treatment modality for sporadic and familial nonampullary nonpolypoid (flat) duodenal adenomas.

DETAILED DESCRIPTION:
Duodenal adenomas are precursors to adenocarcinoma. Treatment with endoscopic polypectomy is technically challenging problematic and associated with a high rate of complication - overall 26%, with bleeding 22-40%, higher with larger polyps. Surgery to remove these benign polyps would be a Whipple operation, which has a high morbidity and 1-4% mortality rate. Medical therapies like celecoxib decrease the number of polyps but do not prevent cancer.

This multicenter prospective cohort study will assess the safety and efficacy of cryoablation treatment as an alternative primary treatment modality for sporadic and familial nonampullary nonpolypoid (flat) duodenal adenomas

Prospective studies have demonstrated the safety and efficacy of nitrous oxide focal cryoballoon ablation for complete eradication of Barrett's esophagus (including a clinical trial published by the Principal Investigator), which is intestinal metaplasia, which is histologically similar to normal duodenal mucosa.

When inflated, the cryoballoon flattens the duodenal folds allowing improved visibility of the duodenal lesions. The focal ablation allows precise targeting and avoidance of the ampulla to minimize pancreatitis risk.

Two cases at Johns Hopkins Hospital have been treated successfully and safely using cryogen dose of 10 seconds. The procedures were easy and short, with excellent views of the lesion with balloon inflation and high definition endoscope. No major adverse events, pain requiring treatment, or bleeding were noted. Minor adverse events included transient abdominal bloating lasting for < 3 days in 1 patient. In one patient with sporadic laterally spreading large Paris 2A polyp who declined standard treatments, complete eradication was achieved with 2 ablation sessions.

In the other patient with familial adenomatous polyposis (FAP) who had 2 hospitalizations for post-polypectomy bleeding after duodenal EMR, complete eradication was noted after 1 treatment of 3 Paris 2A and 2B adjacent polyps.

Follow-up of these two patients shows no recurrence > 1 year and at the most recent follow-up procedures. Clinical and endoscopic surveillance continues.

In addition, another physician at the University of Texas Health Science Center at San Antonio (UTHSCSA) reported another two patients with duodenal adenomas in her practice treated successfully with cryoballoon ablation without complications. Two other collaborating physicians at Memorial Hermann Texas Medical Center in Houston, Texas, and Geisinger Medical Center in Pennsylvania have also reported favorable response of these challenging neoplasms to endoscopic cryoballoon ablation. The group is currently preparing a case series report and a separate Institutional Review Board application is being submitted.

This study may impact on the management of patients with duodenal adenomas by demonstrating the potential for safe and effective non-operative eradication using cryoballoon ablation. The safety profile of endoscopic cryoballoon ablation is likely to be better than endoscopic resection based on a large clinical and research experience in Barrett's esophagus patients (>250) and small clinical experience in duodenal adenoma patients, with <=5% bleeding, no perforation, and transient, mild post-treatment discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic duodenal adenomas between 1 to 5 cm in widest diameter
* FAP patient with Spigelman class 2, 3 or 4 (see definition below)
* Polyp characteristics: Non-polypoid lesions Paris 2A and 2B, or
* Sessile adenomas, occupying no more than 50% circumference of duodenum, and no more than 3 duodenal folds
* Individuals must be considered high risk for surgery or endoscopic resection, due to complication risk, or declined standard therapies.
* Prior endoscopic mucosal resection (EMR) or saline-assisted polypectomy allowed if polyp characteristics meet inclusion criteria.

Exclusion Criteria:

* Suspected or proven duodenal carcinoma
* Paris 1p pedunculated, Paris 2c, or 3 lesions
* Paris 1s lesion > 4 mm thick (estimated with closed biopsy forceps)
* Ampullary lesion or lesion involving the ampulla
* Prior failed ablative treatment with Argon Plasma Coagulation, laser, or cryotherapy
* Pre-existing esophageal, gastric, pyloric, or duodenal stenosis/stricture preventing advancement of a therapeutic endoscope during screening/baseline esophagogastroduodenoscopy (EGD.) Subjects are eligible if the stenosis/stricture is dilated to at least 15mm, but baseline treatment may need to be delayed.
* Any endoscopically-visualized abnormalities such as ulcers, masses or nodules during screening/baseline EGD within 3 cm of the treatment area.
* Subjects with nodular polyps or suspicion of invasive cancer by white light endoscopy /enhanced imaging/biopsy identified during screening/baseline EGD
* Suspicion of malignancy by abdominal or endoscopic ultrasound imaging based on malignant lymph nodes, invasion of lesion beyond mucosa.
* EMR or polypectomy < 6 weeks prior to baseline treatment.
* Untreated invasive esophageal malignancy, including margin-positive EMR.
* Active duodenitis in treatment zone during screening/baseline EGD.
* Severe medical comorbidities precluding endoscopy, or limiting life expectancy to less than 2 years in the judgment of the endoscopist.
* Uncontrolled coagulopathy or inability to be off anticoagulation or anti-platelet medication per standards of the institutions performing cryoablation.
* Known portal hypertension, visible esophageal, gastric, or duodenal varices, or history of varices.
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation.
* Pregnant or planning to become pregnant during period of study participation.
* Patient refuses or is unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety of cryoBalloon ablation in treating non-ampullary non-polypoid duodenal adenomas (DAs) as assessed by the incidence of adverse events in all treated patients | 5 years
  To assess incidence of treatment-related adverse events following cryoablation using the C2 cryoballoon system, defined by frequency or number of adverse events in all treated patients (per patient analysis).
Safety of cryoBalloon ablation in treating non-ampullary non-polypoid duodenal adenomas (DAs) as assessed by the incidence of adverse events in all treatment procedures | 5 years
  To assess incidence of treatment-related adverse events following cryoablation using the C2 cryoballoon system, defined by frequency or number of adverse events in all treatment procedures (per procedure analysis).
Complete eradication rate of DAs | 1 year
  Complete eradication (CE) rate of DAs as assessed by a combination of endoscopic and pathologic absence of adenomatous tissue in treated areas.

SECONDARY OUTCOMES:
Percent change in the treated duodenal adenoma size | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Endoscopic assessment: percent change in adenoma size by blinded review by 3-person expert panel of still images with region of interest marked by tattoo - per lesion analysis and per patient analysis.
Technical failure rate | 5 years
  Technical failure rate is the proportion of treatment procedures with cryoballoon ablation that did not complete delivery of cryogen to all targeted sites.
Change in Spigelman class score | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Percent change in Spigelman classification for polyp burden in FAP patients from baseline to 1 year after treatment is completed. The Spigelman classification assigns points based upon polyp number, polyp size, histology and dysplasia grade, where Stage 0 = 0 points, Stage I = 1-4 points, Stage II = 5-6 points, Stage III = 7-8 points, and Stage IV = 9-12 points. The higher the score, the more severe or advanced the FAP disease in the duodenum.
Progression rate to high grade dysplasia or duodenal cancer | 5 years
  Progression rate: percentage of patients with progression of dysplasia grade to high grade dysplasia or invasive cancer, compared to baseline biopsies, at any time during the study.
Time to complete eradication of DAs in each patient | 5 years
  Time to complete eradication (in months) of all duodenal adenomas in each patient
Time to complete eradication of each treated DA lesion | 5 years
  Time to complete eradication (in months) of each treated DA lesion
Median number of CryoBalloon treatments to complete eradication. | 5 years
  Median number of cryoballoon ablation treatments to achieve complete eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia I. Canto, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Northwell Health, Manhasset, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Submit request to P.I. and study team with study goal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 4 years
Access Criteria: Submit request to P.I. and study team with study goal.